CLINICAL TRIAL: NCT04236505
Title: A Wait List Controlled Trial of Brief ACT and Brief MBSR-informed Group Interventions for Anxiety in a University Setting
Brief Title: Wait List Controlled Trial of Brief ACT and Brief MBSR-informed Group Interventions for Anxiety in a University Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETH1819-0489
Record Dates: First submitted 2019-04-15; First posted 2020-01-22 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Anxiety; Stress
Keywords: Mindfulness; Acceptance and Commitment Therapy (ACT); Student mental health
MeSH Terms: conditions — Anxiety Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Participants are randomised into two intervention groups and a waitlist controlled group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT group intervention (Experimental): 4 weekly 2hour group therapy interventions drawing from an Acceptance and Commitment Therapy (ACT) based protocol.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) group based intervention
- Mindfulness skills group intervention (Experimental): 4 weekly 2 hour group therapy interventions drawing from an Mindfulness based stress reduction (MBSR) based protocol
  Interventions: Behavioral: Mindfulness based stress reduction (MBSR) informed brief mindfulness skills group intervention
- Wait list control group (Placebo Comparator): Wait list control group who at the time of the experimental group interventions are not attending a group and receiving treatment as usual. This group are offered a Mindfulness skills group intervention after the follow up data has been collected.
  Interventions: Behavioral: Wait list Control group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) group based intervention — 4 week ACT psychological intervention group based on Flaxman and McIntosh's ACT in the work place group format
  Arms: ACT group intervention
Behavioral: Mindfulness based stress reduction (MBSR) informed brief mindfulness skills group intervention — 4 week Mindfulness based stress reduction (MBSR) informed brief mindfulness skills group intervention
  Arms: Mindfulness skills group intervention
Behavioral: Wait list Control group — this group are placed on a wait list for group treatment whilst the other experimental groups run. This group are offered the MBSR based mindfulness skills once the follow up data has been collected from the other two experimental groups
  Arms: Wait list control group

SUMMARY:
A randomised wait-list-controlled trial is being run in a psychology department research clinic at a London University providing two four-week group interventions (one Acceptance and Commitment Therapy (ACT) and one MBSR-informed) to students presenting with mild to moderate anxiety. Pre and post measures of anxiety, depression, psychological flexibility, mindfulness, self-compassion, letter-number sequencing and trail making will be collected. Groups will be audio recorded for qualitative analysis and long term follow up outcomes will be collected.

DETAILED DESCRIPTION:
This pilot study is designed as a randomised controlled trial comparing the effectiveness of two group interventions to a waitlist control (WLC) group: The first group is informed by Acceptance and Commitment Therapy (ACT), and the second group is informed by Mindfulness-Based Stress Reduction (MBSR). Student participants in the intervention groups will take part in either four 2-hour group sessions of ACT or MBSR-informed group interventions. Participants who are placed on the waitlist will be offered either brief ACT or brief MBSR-informed groups after 4 weeks. Both intervention and WLC groups will be administered an assessment battery before the interventions start (baseline), and soon after the intervention (post-intervention). All participants will complete the assessment battery measures at 8 weeks after post-measurement (4-week follow-up). After the completion of the 4-week follow-up measures, participants in the WLC group will be randomly allocated to either intervention groups, followed up by a post-measurement 4 weeks later after the completion of each intervention.

METHODS Therapeutic interventions: Participants of the intervention groups will be randomly allocated into either a 4- week ACT or MBSR-informed group. Instructions will be offered by the group facilitators, including discussion, reading assignments, as well as training and practice in a variety of acceptance- and mindfulness-based techniques.

ACT GROUP The ACT protocol proposed in this study has been adapted from a manual developed by Flaxman, McIntosh and Oliver (2018) for ACT training in workplace settings. This protocol has been adapted further by the authors in collaboration with Dr Kornilia Givissi and Dr Hana Villar for use in clinical settings and specifically applied to participants struggling with anxiety. This intervention combines psychoeducational and experiential practices to introduce concepts and develop skills in the six core processes of ACT. Participants will attend 4 two-hour weekly sessions of this group. The first five and last five minutes of each session will be for process measure completion. The focus of each session is detailed in the ACT protocol MBSR-INFORMED GROUP The 4-week MBSR protocol proposed in this study has been adapted from the work of Kabat-Zinn (1990), Segal, Williams, and Teasdale (2002) and has been adapted by Dr Trudi Edginton, an experienced mindfulness teacher. It has synthesised the main elements, includes all of the traditional practices and is congruent with the philosophical underpinning of the original MBSR group. This group consists of 4 two-hour weekly sessions. The first five and last five minutes of each session will be for process measure completion. The focus of each session is detailed in the MBSR-informed protocol .

Waitlist Control (WLC) group: Those assigned to the WLC group will not engage in the group interventions during the course of the intervention period. At the start of the pilot trial, they will be informed of the 4-week waiting period after which they will be randomly allocated into either intervention groups. They will be asked to complete the assessment battery measures at baseline and all follow-up timepoints.

Researcher/Practitioners: The ACT or MBSR-informed protocols in this study will be delivered by qualified and HCPC registered counselling and/or clinical psychology practitioners and are either employed or visiting lecturers in the Department of Psychology. They will all have received training in ACT and/or MBSR, and will undertake weekly clinical peer supervision to ensure fidelity to the intervention models. The research will be evaluated by the named staff members on this application and will not provide interventions but supervision to those delivering the protocols to the study participants.

Evaluation: Evaluation of the study will be conducted by the research clinic team. The evaluation will comprise of the assessment battery measures that will be self- administered at the start of the project and collected by the researcher, and therapy process measures that will be completed at the end of each session. To ensure confidentiality, measures will be de-identified and assigned a code. The researcher will remind the participants that they can choose not to complete the measures or answer any of the questions. Any paper-based measures completed by participants will be stored in a locked filing cabinet in the research clinic office until the data have been entered into a computer, after which hard copies will be securely destroyed. Data collected via tablet or other electronic devices will be stored on a City-protected cloud.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate anxiety

Exclusion Criteria:

* dissociation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire | Measure collected at Baseline (week 0), post treatment (week 6) and at follow up (week 11) in experimental groups and in waiting list control group. .
  The Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011) measures psychological inflexibility or experiential avoidance.This 7-item one-factor scale is scored by adding together the seven items.Higher scores equal greater levels of psychological inflexibility. Measuring change in Psychological Flexibility.
Comprehensive Assessment of Acceptance and Commitment Therapy (CompACT) | Measure collected at baseline (week 0), post each intervention (week 1, 2, 3, 4) and post treatment (week 6) and at follow up (week 11) by experimental group and the waiting list group completed the measure at baseline, post intervention and f-up
  CompACT; Francis, Dawson & Golijani-Moghaddam, 2016) was developed as a general measure of psychological flexibility (and constituent sub-processes) as conceptualized within the ACT model.This 23-item measure has shown initial advantages to the AAQ-II and its inclusion is intended to further test its validity. Measuring change in psychological Psychological flexibility
Five Facet of Mindfulness Questionnaire (FFMQ) - SHORT FORM | Measure collected at baseline (week 0), post each intervention (week 1, 2, 3, 4) and post treatment (week 6) and at follow up (week 11) by experimental group and the waiting list group completed the measure at baseline, post intervention and f-up
  The Five Facet of Mindfulness Questionnaire (FFMQ; Bohlmeijer, Ten Klooster, Fledderus,Veehof,& Baer, 2011) is a 39-item measure consisting of five subscales (1. observing, 2. describing, 3. acting with awareness, 4. non-judging of inner experience, and 5. non-reactivity to inner experience). The FFMQ short-version (24 items) has been used.The FFMQ short-version (24 items) captures 4 of the psychological flexibility processes: contact with the present moment; cognitive defusion; self as context; acceptance.Items of the FFMQ were measured on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true). A global FFMQ score are calculated using the mean of all 24 items (considering reverse-scoring). Measuring changes in mindfulness
Generalised Anxiety Disorder Assessment (GAD-7) | Measure collected at baseline (week 0), post each intervention (week 1, 2, 3, 4) and post treatment (week 6) and at follow up (week 11) by experimental group and the waiting list group completed the measure at baseline, post intervention and f-up
  The Generalised Anxiety Disorder Assessment (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) is used to measure or assess the severity of generalised anxiety disorder (GAD) This self-administered instrument has 7 items. Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day" respectively, and then adding together the scores for the seven questions.
  GAD-7 total score for the seven items ranges from 0 to 21. Scores represent: 0-5 = Mild anxiety, 6-10 = Moderate anxiety, 11-15 = Moderately severe anxiety, and 15-21 = Severe anxiety.
  When used as a screening tool, further evaluation is recommended when the score is 10 or greater. Measuring changes in anxiety scores.
Patient Health Questionnaire-9 (PHQ-9) | Measure collected at baseline (week 0), post each intervention (week 1, 2, 3, 4) and post treatment (week 6) and at follow up (week 11) by experimental group and the waiting list group completed the measure at baseline, post intervention and f-up
  The Patient Health Questionnaire-9 (PHQ-9; Kroenke & Spitzer, 2002) is used to measure or assess the severity of depression.
  This self-administered scale has 9 items. Each item asks the individual to rate the severity of his or her symptoms over the past two weeks.
  Response options include "not at all", "several days", "more than half the days" and "nearly every day" respectively, and then adding together the scores for the seven questions. Scores represent: 5-9 = mild depression / low mood, 0-14 - moderate depression / low mood, 15-19 - moderately severe depression / low mood, and 20-27 - severe depression/low mood. Measuring change in scores of low mood.
  When used as a screening tool, further evaluation is recommended when the score is 10 or greater.

SECONDARY OUTCOMES:
Ruminative Responses Scale | This measure was collected at Baseline (week 0), post treatment (week 6) and at follow up (week 11) in experimental groups and in waiting list control group.
  The Ruminative Responses Scale (RRS) of the Response Styles Questionnaire (RSQ; Nolen-Hoeksema & Morrow, 1991) assesses the extent to which individuals repeatedly focus on the causes, meanings, and consequences of their negative mood.
  This measure has 22 items and a factor analysis of the RRS has identified two separate subscales that are differentially related to symptoms of depression. The first, reflection, consists of five questions that assess the degree to which individuals engage in cognitive problem-solving to improve their. The second, brooding, consists of five items that assess the degree to which individuals passively focus on the reasons for their distress (Treynor et al., 2003).
  Brooding and reflection scores are computed by taking the average of items on each respective scale. Measuring a change in Rumination.
Self compassion scale | Measure collected at Baseline (week 0), post treatment (week 6) and at follow up (week 11) in experimental groups and in waiting list control group.
  This is a measure of self-compassion. This 26-item measure is based on an aggregate of responses on three subscales: (1) self-kindness versus self-judgment, (2) common humanity versus isolation, and (3) mindfulness versus overidentification. Subscale scores are computed by calculating the mean of subscale item responses. To compute a total self-compassion score, reverse score the negative subscale items -self-judgment, isolation, and over-identification (i.e., 1 = 5, 2 = 4, 3 = 3. 4 = 2, 5 = 1) -then compute a total mean. This will measure a change in self compassion.
student engagement scale | Measure collected at Baseline (week 0), post treatment (week 6) and at follow up (week 11) in experimental groups and in waiting list control group.
  Student Engagement Scale (SES; Gunuc & Kuzu, 2015) is a measure of student engagement for higher education. This 41-item measure consists of six subscales: 1) valuing, 2) sense of belonging, 3) cognitive engagement, 4) peer relationships (emotional engagement-I), 5) relationships with faculty members (emotional engagement-II), and 6) behavioural engagement.
  Items of the SES are measured on a five-point Likert-type scale ranging from 1 (I totally disagree) to 5 (I totally agree).
  Higher student engagement scores indicate that the student has a high level of engagement with the university, campus and class.
  This will measure a change in student engagement.
Trail making test | Measure collected at Baseline (week 0), post treatment (week 6) and at follow up (week 11) in experimental groups and in waiting list control group.
  Trail Making Test (TMT; Arnett, Seth & Labovitz, 1995) is a neuropsychological test of visual attention and task switching.The standard TMT comes in two forms: Trails A, where subjects connect a series of 25 numbered circles in ascending order, and Trails B, where subjects connect 25 circles alternating between ascending numbers and letters (e.g., 1-A-2-B, etc.).Completion times (in seconds) on the TMT are used to assess visual attention, speed of processing, mental flexibility, and executive function in patients by comparisons with normative data from appropriate control populations (Tombaugh, 2004). Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
WAIS-1V Letter-number sequencing | Measure collected at Baseline (week 0), post treatment (week 6) and at follow up (week 11) in experimental groups and in waiting list control group.
  WAIS-IV subtest Letter-Number Sequencing (LNS) is a well-validated measure of manipulation WM (Snyder, Miyake, & Hankin, 2015). The participant is read a series of numbers and letters and asked to recall the numbers in ascending order, followed by the letters in alphabetical order.The number of items is 21. With each item being marked 0 if reported incorrectly or 1 if reported correctly, the maximum score is 21. This is to measure the change in letter-number sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychology Department, City, University of London, London, United Kingdom